CLINICAL TRIAL: NCT06902467
Title: Combined Intraperitoneal Chemotherapy Regimen After Optimal Interval Surgery in Advanced Ovarian Cancer: BICOV-1 (Bidirectional Chemotherapy in Ovarian Cancer)
Acronym: BICOV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMIB-BICOV-2022-01
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Following 3 or 4 cycles of systemic neoadjuvant chemotherapy and complete interval CC-0 surgery, patients in the study will receive 4 cycles of 21 days every 3 weeks of the regimen studied by Armstrong 8 and modified by GEICO 18: IV paclitaxel 175 mg /m2 (day 1) + IP cisplatin 100 mg/m2 (day 2) + IP paclitaxel 60 mg/m2 (day 8).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Following 3 or 4 cycles of systemic neoadjuvant chemotherapy and complete interval CC-0 surgery, pat (Experimental): Following 3 or 4 cycles of systemic neoadjuvant chemotherapy and complete interval CC-0 surgery, patients in the study will receive 4 cycles of 21 days every 3 weeks of the regimen studied by Armstrong 8 and modified by GEICO 18: IV paclitaxel 175 mg /m2 (day 1) + IP cisplatin 100 mg/m2 (day 2) + IP paclitaxel 60 mg/m2 (day 8).
  Interventions: Drug: Following 3 or 4 cycles of systemic neoadjuvant chemotherapy and complete interval CC-0 surgery, patients in the study will receive 4 cycles of 21 days every 3 weeks of the regimen studied by Armstron

INTERVENTIONS:
Drug: Following 3 or 4 cycles of systemic neoadjuvant chemotherapy and complete interval CC-0 surgery, patients in the study will receive 4 cycles of 21 days every 3 weeks of the regimen studied by Armstron — Following 3 or 4 cycles of systemic neoadjuvant chemotherapy and complete interval CC-0 surgery, patients in the study will receive 4 cycles of 21 days every 3 weeks of the regimen studied by Armstrong 8 and modified by GEICO 18: IV paclitaxel 175 mg /m2 (day 1) + IP cisplatin 100 mg/m2 (day 2) + IP paclitaxel 60 mg/m2 (day 8).

SUMMARY:
A multicenter, low-intervention, drug-based study to evaluate the feasibility and safety of a combined regimen of two intraperitoneal chemotherapy modalities (used in routine clinical practice) following interval surgery for the treatment of advanced ovarian cancer. This is an independent research project (free of commercial interests).

DETAILED DESCRIPTION:
Based on the available evidence, an optimized protocol is proposed for the radical approach to primary advanced ovarian cancer with peritoneal dissemination (FIGO III/IV). After optimal interval surgery defined as CRS + HIPEC, bidirectional therapy (BIC) will be evaluated, reproducing the scheme studied by Armstrong 8 with the modifications and recommendations of GEICO (Spanish Ovarian Cancer Research Group) 18. A series of measures are proposed to minimize the risk of complications and toxicity related to intraperitoneal treatment. All of this, with the ultimate objective of maximizing the patient's disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-70 years with a histologically proven diagnosis of FIGO stage IIIB-C/IV epithelial ovarian cancer (high-grade serous epithelial carcinoma)
* Absence of extraperitoneal disease.
* Good performance status: Karnofsky score >70 or Performance status <= 2
* Adequate liver function, defined as bilirubin <0.15 times the upper limit of normal (ULN), aspartate aminotransferase and alanine aminotransferase <= 2.5 times ULN, and alkaline phosphatase <= 3 times ULN.
* Adequate renal function, defined as serum creatinine <= 1.5 times ULN
* Acceptable bone marrow function, defined as neutrophils >1.5 x 106 L-1, hemoglobin >10 g/dL-1, and platelets >100.0 x 109 L-1
* Absence of cardiac, pulmonary, hepatic, renal, or neurological disease that contraindicates major surgery.
* Negative serum and urine pregnancy test results for women of childbearing potential at the screening visit.
* Administration of neoadjuvant chemotherapy with a total of 3 or 4 systemic cycles.
* Surgery with complete CC0 cytoreduction without digestive anastomoses.
* Patients who have signed the written IC.

Exclusion Criteria:

* Disease progression during systemic treatment with neoadjuvant chemotherapy.
* Extraperitoneal disease (including retroperitoneal lymph node metastases)
* Inability to achieve complete cytoreduction (CC-0) during preoperative (imaging) or intraoperative evaluation.
* Performance of at least one digestive anastomosis of any type. Active infection of any origin
* Allogeneic transplant, or prior bone marrow transplant, or high-dose chemotherapy with bone marrow or stem cell rescue.
* Participation in a clinical trial with an investigational drug within the last 30 days.
* Pregnant or breastfeeding women, where pregnancy is defined as the state of a woman after conception and until the end of pregnancy, confirmed by a positive human chorionic gonadotropin (hCG) test result, or who plan to become pregnant or breastfeed during study treatment or within 30 days of the end of treatment with the study drug.
* Patients with a history of allergic reactions or hypersensitivity to drugs chemically related to cisplatin and paclitaxel.
* Failure to sign written informed consent.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Twenty patients aged between 18 and 75 years, diagnosed with FIGO stage IIIB-IV epithelial ovarian cancer (high-grade serous epithelial carcinoma) and previously treated with systemic neoadjuvant chemotherapy, followed by cytoreduction + HIPEC and postoperative combined systemic and intraperitoneal chemotherapy, will be initially selected.
Enrollment: 20 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Disease-free interval | Up to 5 years
  Number of days without disease

SECONDARY OUTCOMES:
Safety related to the intervention | Up to 5 years
  Number of adverse events reported
Quality of life of the participants | Up to 5 years
  To evaluate the Quality of Life parameters of patients before surgery, before the start of treatment and after its completion (3 and 6 months).
  EQ-5D SCALE, 20-centimeter vertical EVA, measured in millimeters, ranging from 0 (worst imaginable health condition) to 100 (best imaginable health condition).

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Cascales Campos, MD, Principal Investigator — HCUVA
Locations (1):
- HCUVA, Murcia, Spain